CLINICAL TRIAL: NCT02726581
Title: An Open-Label, Randomized Phase 3 Trial of Combinations of Nivolumab, Pomalidomide and Dexamethasone in Relapsed and Refractory Multiple Myeloma
Brief Title: An Investigational Immuno-therapy Study of Nivolumab, Pomalidomide and Dexamethasone Combinations in Patients With Multiple Myeloma
Acronym: CheckMate 602
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-602; 2015-005699-21 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-04-01 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Nivolumab; elotuzumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational Arm (Experimental): Nivolumab, Pomalidomide and Dexamethasone
  Enrollment is closed for this arm
  Interventions: Biological: Nivolumab; Drug: Pomalidomide; Drug: Dexamethasone
- Control Arm (Active Comparator): Pomalidomide and Dexamethasone
  Enrollment is closed for this arm
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Exploratory Arm (Experimental): Nivolumab, Elotuzumab, Pomalidomide and Dexamethasone
  Enrollment is closed for this arm
  Interventions: Biological: Nivolumab; Biological: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days, IV (intravenous)
  Other Names: BMS-936558
  Arms: Exploratory Arm; Investigational Arm
Biological: Elotuzumab — Specified dose on specified days, IV
  Other Names: BMS-901608
  Arms: Exploratory Arm
Drug: Pomalidomide — Specified dose on specified days, PO (by mouth)
Drug: Dexamethasone — Specified dose on specified days, PO

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of several combination therapies for Multiple Myeloma. Upon entry into the study, patients will be randomized (assigned by chance) to receive either:

Group 1: nivolumab, pomalidomide and dexamethasone OR Group 2: pomalidomide and dexamethasone OR Group 3: nivolumab, elotuzumab, pomalidomide and dexamethasone.

Enrollment is closed for all groups.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed and refractory multiple myeloma
* Measurable disease
* Have received ≥ 2 lines of prior therapy which must have included an immune modulatory drug (IMiD) and a proteasome inhibitor alone or in combination

Exclusion Criteria:

* Solitary bone or extramedullary plasmacytoma disease only
* Active plasma cell leukemia

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (121):
- United States (72):
  - Local Institution - 0020, Birmingham, Alabama
  - Local Institution - 0160, Mobile, Alabama
  - Local Institution - 0163, Fayetteville, Arkansas
  - Local Institution - 0118, Bakersfield, California
  - Local Institution - 0093, Corona, California
  - Local Institution - 0016, Fountain Valley, California
  - Local Institution - 0164, La Jolla, California
  - UC San Diego Moores Cancer Ctr, La Jolla, California
  - Local Institution - 0138, Los Angeles, California
  - Local Institution - 0155, Los Angeles, California
  - Local Institution - 0117, Redondo Beach, California
  - Local Institution - 0092, Riverside, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Local Institution - 0113, Santa Maria, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Poudre Valley Health Care, Fort Collins, Colorado
  - Local Institution - 0116, Grand Junction, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Local Institution - 0147, Washington D.C., District of Columbia
  - Local Institution - 0011, Boynton Beach, Florida
  - Florida Cancer Specialists S., Fort Myers, Florida
  - Local Institution - 0114, Hollywood, Florida
  - Cancer Specialists of North FL, Jacksonville, Florida
  - Local Institution - 0082, Pensacola, Florida
  - Local Institution - 0126, St. Petersburg, Florida
  - Local Institution - 0130, Tallahassee, Florida
  - Local Institution - 0125, West Palm Beach, Florida
  - Local Institution - 0119, Athens, Georgia
  - Local Institution - 0009, Atlanta, Georgia
  - Local Institution - 0024, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Local Institution - 0035, Chicago, Illinois
  - Local Institution - 0111, Fort Wayne, Indiana
  - Indiana University Cancer Ctr, Indianapolis, Indiana
  - Local Institution - 0018, Bethesda, Maryland
  - Local Institution - 0006, Baltimore, Massachusetts
  - Local Institution - 0123, Worcester, Massachusetts
  - Local Institution - 0150, Ypsilanti, Michigan
  - Local Institution - 0137, Hattiesburg, Mississippi
  - St. Louis Cancer Care, Llp, Bridgeton, Missouri
  - Local Institution - 0128, Kansas City, Missouri
  - Local Institution - 0049, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - Local Institution - 0079, Lincoln, Nebraska
  - Local Institution - 0076, Flemington, New Jersey
  - Local Institution - 0002, Hackensack, New Jersey
  - Local Institution - 0095, New Brunswick, New Jersey
  - Local Institution - 0142, Paramus, New Jersey
  - Local Institution - 0010, Buffalo, New York
  - Broome Oncology LLC, Johnson City, New York
  - Mount Sinai Medical Center, New York, New York
  - Local Institution - 0017, New York, New York
  - Local Institution - 0001, Durham, North Carolina
  - Local Institution - 0096, Winston-Salem, North Carolina
  - Local Institution - 0012, Columbus, Ohio
  - University Of Oklahoma, Oklahoma City, Oklahoma
  - Local Institution - 0145, Portland, Oregon
  - Local Institution - 0136, Lancaster, Pennsylvania
  - Local Institution - 0021, Philadelphia, Pennsylvania
  - Local Institution - 0036, Sayre, Pennsylvania
  - Local Institution - 0152, Greenville, South Carolina
  - Local Institution - 0069, Germantown, Tennessee
  - Tennessee Oncology, PLLC - SCRI - PPDS, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Local Institution - 0044, Houston, Texas
  - Local Institution - 0037, San Antonio, Texas
  - Local Institution - 0046, Temple, Texas
  - Local Institution - 0022, Ogden, Utah
  - Local Institution - 0153, Salt Lake City, Utah
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Local Institution - 0144, Seattle, Washington
- Austria (5):
  - Local Institution - 0029, Linz
  - Universitaetsklinik Salzburg, Salzburg
  - Local Institution - 0026, Vienna
  - Wilhelminenspital, Vienna
  - Klinikum Wels-Grieskirchen Gmbh, Wels
- Canada (8):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution - 0074, Toronto, Ontario
  - Local Institution - 0039, Montreal, Quebec
  - MUHC - Glen Site, Montreal, Quebec
  - Local Institution - 0154, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution - 0157, Rimouski, Quebec
- Czechia (3):
  - Interni hematologicka a onkologicka klinika, Brno
  - Klinika hematoonkologie, Ostrava-Poruba
  - I. interni klinika - klinika hematologie 1. LF UK a VFN v Praze, Prague
- Denmark (2):
  - Local Institution, Aarhus
  - Local Institution, Odense
- Germany (6):
  - Local Institution - 0050, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Uniklinikum Duesseldorf, Düsseldorf
  - Local Institution - 0135, Kiel
  - Klinikum Der Johannes Gutenberg Universitaet Mainz, Mainz
  - Local Institution - 0054, Ulm
- Alexandra General Hospital Of Athens, Athens, Greece
- Israel (5):
  - Local Institution - 0087, Beersheba
  - Local Institution, Jerusalem
  - Local Institution, Petah Tikva
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (6):
  - Local Institution - 0042, Turin, Piedmont
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Di Ancona, Ancona
  - Local Institution - 0089, Bergamo
  - A. O. U. Di Bologna, Policlinico S. Orsola Malpighi, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola (FC)
  - Azienda Ospedaliera Santa Maria Terni, Terni
- Norway (2):
  - Local Institution, Oslo
  - Local Institution - 0075, Stavanger
- Portugal (2):
  - Local Institution - 0132, Lisbon, Lisbon District
  - Local Institution, Porto
- Local Institution - 0071, San Juan, Puerto Rico
- Spain (5):
  - Local Institution - 0101, Pozuelo de Alarcón, Madrid
  - Local Institution - 0098, Badalona-Barcelona
  - Local Institution - 0100, Barcelona
  - Local Institution - 0097, Pamplona
  - Local Institution - 0099, Salamanca
- Local Institution - 0064, Huddinge, Sweden
- Hopitaux Universitaires de Geneve, Geneva, Switzerland
- Local Institution - 0186, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study contains an exploratory third arm evaluating the clinical benefit and the safety of the combination therapy of elotuzumab, nivolumab, pomalidomide and dexamethasone (Arm C: NE-Pd). Participants randomized to the Pd arm were allowed to cross over to this exploratory NE-Pd arm at the time of progression.
Groups:
- Arm A: N-Pd: Nivolumab:
  * Cycles 1 through 4: 240 mg IV Days 1, 15 of each 28-day cycle.
  * Cycles 5 and beyond: 480 mg IV Day 1 of each 28-day cycle.
  Pomalidomide:
  - 4 mg PO QD Days 1-21 of each 28-day cycle.
  Dexamethasone:
  * Participants </= 75 years old: 40 mg PO Days (1, 8, 15, and 22) of each cycle
  * Participants > 75 years old: 20 mg PO Days (1, 8, 15, and 22) of each cycle.
- Arm B: Pd: Pomalidomide:
  - 4 mg PO QD Days 1-21 of each 28-day cycle.
  Dexamethasone:
  * Participants </= 75 years old: 40 mg PO Days (1, 8, 15, and 22) of each cycle
  * Participants > 75 years old: 20 mg PO Days (1, 8, 15, and 22) of each cycle.
- Arm C: NE-Pd: Nivolumab:
  * Cycles 1 through 4: 240 mg IV Days 1, 15 of each 28-day cycle.
  * Cycles 5 and beyond: 480 mg IV Day 1 of each 28-day cycle.
  Elotuzumab:
  * Cycles 1 - 2: 10 mg/kg IV Days 1, 8, 15, and 22 of each 28-day cycle.
  * Cycle 3 and 4: 10mg/kg IV Day 1 and 15 of each 28-day cycle.
  * Cycles 5 and beyond: 20 mg/kg IV Day 1 of each 28-day cycle.
  Pomalidomide:
  4 mg PO QD Days 1-21 of each 28-day cycle.
  Dexamethasone:
  Days 1, 8, 15, and 22 of each cycle.
  * Participants </= 75 years old: weeks with elotuzumab dosing: 28 mg PO + 8 mg IV and 40 mg PO on non-elotuzumab dosing weeks.
  * Participants > 75 years old: weeks with elotuzumab dosing: 8 mg PO + 8 mg IV and 20 mg PO on non-elotuzumab dosing weeks.
Period: Pre-Treatment Period
Arm/Group | Arm A: N-Pd | Arm B: Pd | Arm C: NE-Pd
Started | 75 | 71 | 24
Completed | 72 | 70 | 24
Not Completed | 3 | 1 | 0
Not completed — Participant request to discontinue study treatment | 0 | 1 | 0
Not completed — Administrative reason by sponsor | 2 | 0 | 0
Not completed — Participant no longer meets study criteria | 1 | 0 | 0
Period: Treatment Period
Arm/Group | Arm A: N-Pd | Arm B: Pd | Arm C: NE-Pd
Started | 72 | 70 | 24
NE-Pd Crossover | 0 | 8 | 0
Completed (Completed treatment) | 0 | 0 | 0
Not Completed | 72 | 70 | 24
Not completed — Disease progression | 47 | 50 | 16
Not completed — Other reasons | 9 | 8 | 2
Not completed — Study drug toxicity | 6 | 3 | 2
Not completed — Adverse event unrelated to study drug | 4 | 4 | 2
Not completed — Participant withdrew consent | 3 | 1 | 1
Not completed — Participant request to discontinue study treatment | 1 | 1 | 1
Not completed — Maximum clinical benefit | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Poor/non-compliance | 1 | 0 | 0
Not completed — Participant no longer meets study criteria | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: N-Pd | Arm B: Pd | Arm C: NE-Pd | Total
Number analyzed (Participants) | 75 | 71 | 24 | 170
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (9.4) | 65.5 (8.7) | 66.2 (11.5) | 65.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 8 | 57
  Male | 51 | 46 | 16 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 6
  Not Hispanic or Latino | 40 | 41 | 15 | 96
  Unknown or Not Reported | 34 | 26 | 8 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 5 | 13
  White | 72 | 64 | 19 | 155
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Randomization to first documented tumor progression or death due to any cause, whichever occurred first. Participants who die without reported prior progression are considered to have progressed on date of their death. Participants who did not progress or die will be censored at their last efficacy assessment. Participants who did not have on study efficacy assessments and alive will be censored on randomization date. Participants who started subsequent anti-cancer therapy without prior reported progression will be censored at last efficacy assessment prior to subsequent anti-cancer therapy. Progression is 1) increase of 25% from lowest confirmed response value in specific Serum M-protein and Urine M-protein criteria and increase of FLC for patients with no measurable M protein in blood or urine at baseline and/or 2) appearance of a new lesion(s), >/= 50% increase from nadir in SPD of > 1 lesion, or >/= 50% increase in the longest diameter of a previous lesion > 1 cm in short axis.
Time Frame: From randomization to the date of the first documented tumor progression or death due to any cause, whichever occurred first (Up to approximately 64 month)
Population: All randomized participants in Arm A and B. Data was pre-specified to be collected only in the N-Pd and Pd arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: N-Pd | Arm B: Pd
Number analyzed (Participants) | 75 | 71
Months | 8.38 [5.78 to 12.06] | 7.33 [6.47 to 8.44]
Statistical Analysis 1: Comparison: Arm A: N-Pd vs Arm B: Pd; Test type: Superiority; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.62 to 1.30]

2. Secondary Outcome: Overall Survival (OS)
Description: The time between the date of randomization and the date of death due to any cause. OS will be censored on the last date a participant was known to be alive.
Time Frame: From randomization to the date of death due to any cause (up to approximately 64 months)
Population: All randomized participants in Arm A and B. Data was pre-specified to be collected only in the N-Pd and Pd arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: N-Pd | Arm B: Pd
Number analyzed (Participants) | 75 | 71
Months | 24.87 [15.61 to 34.40] | 21.39 [17.91 to 27.56]
Statistical Analysis 1: Comparison: Arm A: N-Pd vs Arm B: Pd; Test type: Superiority; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.53 to 1.19]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of randomized participants who achieved a best overall response (BOR) of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) using International Myeloma Working Group (IMWG) criteria.
  sCR= Complete response as defined below plus normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry.
  CR = Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates.
  VGPR = Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >/= 90% reduction in serum M-protein plus urine M-protein level < 100 mg per 24 h.
  PR = >/= 50% reduction of serum M-protein plus reduction in 24 h urinary M-protein by >/= 90% or to < 200 mg per 24 h.
Time Frame: From randomization up to approximately 64 months
Population: All randomized participants in Arm A and B. Data was pre-specified to be collected only in the N-Pd and Pd arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: N-Pd | Arm B: Pd
Number analyzed (Participants) | 75 | 71
Percentage of participants | 48.0 [36.3 to 59.8] | 54.9 [42.7 to 66.8]
Statistical Analysis 1: Comparison: Arm A: N-Pd vs Arm B: Pd; Test type: Superiority; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.39 to 1.46]

4. Secondary Outcome: Time to Objective Response (TTR)
Description: The time from the date of randomization to the date of the first stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR= Complete response as defined below plus normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry.
  CR = Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates.
  VGPR = Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >/= 90% reduction in serum M-protein plus urine M-protein level < 100 mg per 24 h.
  PR = >/= 50% reduction of serum M-protein plus reduction in 24 h urinary M-protein by >/= 90% or to < 200 mg per 24 h.
Time Frame: From the date of randomization to the date of the first sCR, CR, VGPR, or PR (up to approximately 64 months)
Population: All responders (sCR, CR, VGPR, or PR) in Arm A and B. Data was pre-specified to be collected only in the N-Pd and Pd arms.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Arm A: N-Pd | Arm B: Pd
Number analyzed (Participants) | 36 | 39
Months | 5.91 (9.09) | 4.37 (5.63)

5. Secondary Outcome: Duration of Objective Response (DOR)
Description: The time between the date of first response to the date of the first objectively documented tumor progression as assessed by the investigator according to International Myeloma Working Group (IMWG) criteria or death due to any cause prior to subsequent anti-cancer therapy. Participants who neither progress nor die will be censored on the date of their last tumor assessment prior to subsequent anti-cancer therapy. Progression is 1) increase of 25% from lowest confirmed response value in specific Serum M-protein and Urine M-protein criteria and increase of FLC for patients with no measurable M protein in blood or urine at baseline and/or 2) appearance of a new lesion(s), >/= 50% increase from nadir in SPD of > 1 lesion, or >/= 50% increase in the longest diameter of a previous lesion > 1 cm in short axis.
Time Frame: From randomization to the date of the first objectively documented tumor progression or death due to any cause prior to subsequent anti-cancer therapy (up to approximately 64 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: N-Pd | Arm B: Pd
Number analyzed (Participants) | 36 | 39
Months | 8.51 [6.47 to 13.83] | 6.47 [5.55 to 11.07]

ADVERSE EVENTS:
Time Frame: AEs and SAEs assessed from first dose to 100 days post last dose (up to approximately 63 months). Participants were assessed for all-cause mortality from their randomization to the study's Primary completion (up to approximately 64 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Arm B: NE-Pd Crossover: Participants who progressed on the Pd control arm and were allowed to crossover to the NE-Pd exploratory arm.
Arm/Group | Arm A: N-Pd | Arm B: Pd | Arm C: NE-Pd | Arm B: NE-Pd Crossover
All-Cause Mortality (participants affected / at risk) | 47/75 | 49/71 | 17/24 | 5/8
Serious Adverse Events (participants affected / at risk) | 52/72 | 41/70 | 18/24 | 5/8
Other Adverse Events (participants affected / at risk) | 70/72 | 65/70 | 24/24 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: N-Pd (N=72) | Arm B: Pd (N=70) | Arm C: NE-Pd (N=24) | Arm B: NE-Pd Crossover (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Condition aggravated (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 4 | 1 | 0
Sudden death (General disorders) | 2 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 3 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 17 | 6 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 8 | 3 | 3 | 1
Septic shock (Infections and infestations) | 0 | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 6 | 4 | 2
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 3 | 4 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: N-Pd (N=72) | Arm B: Pd (N=70) | Arm C: NE-Pd (N=24) | Arm B: NE-Pd Crossover (N=8)
Anaemia (Blood and lymphatic system disorders) | 26 | 20 | 11 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 24 | 22 | 10 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 11 | 4 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 2 | 0
Hypothyroidism (Endocrine disorders) | 4 | 0 | 2 | 0
Cataract (Eye disorders) | 4 | 4 | 0 | 0
Vision blurred (Eye disorders) | 10 | 2 | 1 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 5 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 17 | 15 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 22 | 17 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 14 | 11 | 4 | 2
Vomiting (Gastrointestinal disorders) | 5 | 6 | 2 | 1
Asthenia (General disorders) | 15 | 12 | 4 | 2
Chest pain (General disorders) | 3 | 4 | 0 | 0
Chills (General disorders) | 2 | 4 | 0 | 1
Fatigue (General disorders) | 34 | 24 | 10 | 6
Non-cardiac chest pain (General disorders) | 5 | 4 | 0 | 0
Oedema peripheral (General disorders) | 14 | 15 | 7 | 1
Pain (General disorders) | 1 | 6 | 1 | 1
Pyrexia (General disorders) | 10 | 9 | 14 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 8 | 5 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 3 | 3 | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 12 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 10 | 12 | 5 | 0
Respiratory tract infection (Infections and infestations) | 9 | 6 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 22 | 3 | 0
Urinary tract infection (Infections and infestations) | 7 | 5 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 4 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 2 | 0
Blood creatinine increased (Investigations) | 8 | 4 | 3 | 0
Lymphocyte count decreased (Investigations) | 7 | 6 | 1 | 0
Neutrophil count decreased (Investigations) | 7 | 6 | 3 | 0
Platelet count decreased (Investigations) | 5 | 7 | 4 | 1
Weight decreased (Investigations) | 4 | 0 | 3 | 2
White blood cell count decreased (Investigations) | 6 | 7 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 10 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 3 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 10 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 3 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 6 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 7 | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 4 | 1 | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 8 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 15 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 11 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 4 | 5 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2 | 1
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 8 | 10 | 7 | 0
Headache (Nervous system disorders) | 7 | 7 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 6 | 2 | 1
Paraesthesia (Nervous system disorders) | 3 | 4 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 1 | 1 | 0
Tremor (Nervous system disorders) | 8 | 6 | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 4 | 2 | 0
Confusional state (Psychiatric disorders) | 5 | 6 | 2 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 11 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 4 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | 6 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 15 | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 4 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 8 | 3 | 1
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 4 | 9 | 2 | 0
Hypotension (Vascular disorders) | 3 | 1 | 3 | 1

LIMITATIONS AND CAVEATS:
Due to the early enrolment termination to Study CA209602 and the smaller than planned study sample size, the statistical analyses were not sufficiently powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT02726581/Prot_SAP_000.pdf